CLINICAL TRIAL: NCT00958035
Title: Study of Bimatoprost Solution in Increasing Eyelash Prominence in African Americans With Eyelash Hypotrichosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 192024-039
Record Dates: First submitted 2009-08-11; First posted 2009-08-13 (Estimated); Results first posted 2012-01-05 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2011-11

CONDITIONS: Hypotrichosis
MeSH Terms: conditions — Hypotrichosis | interventions — Solutions; Bimatoprost

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- LATISSE® (Experimental): bimatoprost ophthalmic 0.03% solution
  Interventions: Drug: bimatoprost ophthalmic 0.03% solution
- Placebo (Placebo Comparator): vehicle sterile solution
  Interventions: Drug: vehicle sterile solution (placebo)

INTERVENTIONS:
Drug: bimatoprost ophthalmic 0.03% solution — Apply one drop of study medication along the upper eyelid margin once daily in the evening
  Other Names: LATISSE®
  Arms: LATISSE®
Drug: vehicle sterile solution (placebo) — Apply one drop of study medication along the upper eyelid margin once daily in the evening
  Arms: Placebo

SUMMARY:
This study will evaluate the safety and efficacy of bimatoprost solution 0.03% once daily to the upper eyelid margins (where the eyelashes meet the skin) compared with vehicle in increasing overall eyelash prominence in self-identified African American/ethnic black subjects exhibiting hypotrichosis of the eyelashes (inadequate or not enough eyelashes).

ELIGIBILITY:
Inclusion Criteria:

* African American/ethnic black
* Adults at least 18 years of age
* Eyelash prominence assessment of minimal or moderate

Exclusion Criteria:

* Subjects with uneven lashes or longer on one side than the other
* Any eye disease or abnormality
* Eye surgery
* Severe hyperpigmentation around the eye
* Eyelash implants
* Eyelash extension application
* Any use of eyelash growth products within 6 months
* Any use of prescription eyelash growth products
* Treatments that may affect hair growth
* Requiring eye drop medications for glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2009-11; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LATISSE® | Placebo
Started | 46 | 43
Completed | 43 | 39
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LATISSE® | Placebo | Total
Number analyzed (Participants) | 46 | 43 | 89
Age, Customized [Number; unit: participants]
  < 45 years | 19 | 16 | 35
  45 - 65 years | 25 | 25 | 50
  > 65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 42 | 88
  Male | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Treatment Responders in Overall Eyelash Prominence at Month 4
Description: Percentage of treatment responders in overall eyelash prominence, defined as at least a 1-grade improvement from baseline at Month 4 in the Global Eyelash Assessment (GEA) Scale. The GEA is a 4-point scale in which eyelash prominence is assessed from 1 (minimal prominence) to 4 (very marked prominence).
Time Frame: Month 4
Population: Intent-to-Treat: All randomized subjects
Measure: Number; unit: Percentage of Patients
Arm/Group | LATISSE® | Placebo
Number analyzed (Participants) | 46 | 43
Percentage of Patients | 69.6 | 48.8

ADVERSE EVENTS:
Arm/Group | LATISSE® | Placebo
Serious Adverse Events (participants affected / at risk) | 1/46 | 1/43
Other Adverse Events (participants affected / at risk) | 14/46 | 4/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LATISSE® (N=46) | Placebo (N=43)
Hepatic Failure (Hepatobiliary disorders) | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LATISSE® (N=46) | Placebo (N=43)
Eyelids Pruritus (Eye disorders) | 3 | 3
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 11 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo